CLINICAL TRIAL: NCT00723476
Title: Family Centered Advanced Care Planning (FCACP)
Brief Title: Family Centered Advanced Care Planning for Adolescents With HIV/AIDS and Their Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maureen Lyon (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor-Investigator, Maureen Lyon, Clinical Health Psychologist, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R34MH072541 (NIH); R34MH072541 (NIH)
Record Dates: First submitted 2008-07-25; First posted 2008-07-28 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: HIV Infections
Keywords: Quality of Life; Adolescent; Advance Care Planning; Palliative Care; End-of-Life Care; HIV/AIDS; Psychological Adjustment
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Participants will receive three 60- to 90-minute health education control sessions.
  Interventions: Behavioral: Health education control sessions
- B (Experimental): Participants will receive three 60- to 90-minute Family Centered Advanced Care Planning sessions.
  Interventions: Behavioral: Family Centered Advanced Care Planning (FCACP) sessions

INTERVENTIONS:
Behavioral: Family Centered Advanced Care Planning (FCACP) sessions — FCACP will include three 60- to 90-minute weekly sessions. Sessions consisting of structured conversations with HIV infected adolescents, their proxies, and trained facilitators will aim to enhance quality of life by integrating effective end-of-life (EOL) care and minimizing depression and anxiety. The three sessions will consist of a structured EOL survey, an FCACP interview, and a family problem-solving lesson.
  Arms: B
Behavioral: Health education control sessions — Health education control sessions will include three 60- to 90-minute sessions and will involve adolescents with HIV/AIDS and their proxies. Topics covered during sessions will include developmental history, planning for the future, and safety tips.
  Arms: A

SUMMARY:
This study will examine the efficacy of Family Centered Advance Care Planning in enhancing quality of life, integrating effective end-of-life care, and preventing depression and anxiety among HIV infected adolescents and their family members.

DETAILED DESCRIPTION:
More than 30,000 adolescents in the United States die annually from the effects of chronic illnesses. The anxiety from facing a terminal illness often hinders adolescents in making decisions about their own end-of-life (EOL) care. Although minors' preferences are not legally binding, legislature, research, and professional guidelines all recommend that adolescent patients become involved in EOL decisions as part of routine intervention while they are stable. Family Centered Advance Care Planning (FCACP) is an intervention that facilitates EOL discussion among adolescents, their families, and their care providers. This pilot study will examine FCACP's effects on adaptive coping, psychological adjustment, quality of life, and plans and actions in HIV infected adolescents. The study will also provide feedback used for improving the FCACP Web site.

This study will include HIV or AIDS infected adolescents ranging in age from 14 to 21 who will jointly enroll with a selected surrogate older than 21. The adolescent/surrogate pairs will be randomly assigned to receive either the FCACP intervention or a health education control intervention. Pairs not immediately ready to participate will form an observational group. Pairs in the FCACP group will meet with a trained facilitator weekly for a 60- to 90-minute session for a total of 3 weeks. During the first session, participants will take the Lyon Advance Care Planning Survey. The second session will consist of the Respecting Choices Interview, where patients will discuss treatment preferences. The Family Problem-Solving session will be last, culminating with the patient's completion of an advance directive. The control groups will follow the same meeting schedule, but will receive health education sessions, not FCACP sessions. Standardized self-report measures will be administered upon entry, after completion of the sessions, and at a 3-month follow up. Usage data will also be analyzed regarding feasibility and acceptability of FCACP as a standard treatment.

ELIGIBILITY:
Inclusion Criteria:

Adolescent Eligibility Criteria:

* Diagnosed with HIV/AIDS
* Between the ages of 14 and 21 years
* Aware of his or her HIV status
* Able to speak English
* Intelligence Quotient (IQ) greater than 69 (all patients have IQ testing results in chart as part of standard of care)
* Consent from the legal guardian if between ages of 14 and 17
* Consent from the surrogate if between ages of 18 and 21
* Assent from adolescent aged 14 to 17
* Consent from adolescent aged 18 to 21

Legal Guardian Eligibility Criteria (for guardians of adolescents aged 14 to 17):

* Adolescent is willing to discuss problems related to HIV with him/her
* Age 21 or older
* Able to speak English
* Legal guardian

Surrogate Eligibility Criteria:

* Selected by adolescent aged 18 to 21
* Age 21 or older
* Willing to discuss problems related to HIV and EOL
* Able to speak English

Exclusion Criteria For All Participants:

* Depression in the moderate to severe range on Beck Depression Inventory
* Unaware of HIV status of self, or if proxy, of adolescent
* Presence of HIV dementia, determined at screening using the HIV Dementia Scale
* Active homicidality or suicidality, determined at baseline screening by psychologist or researcher

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2005-09; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Improved mental health outcomes (e.g., decreased anxiety, depression), improved quality of life, and improved plans and actions (e.g., communication with primary health care provider, an advanced directive in the medical chart) | Measured at Month 3 of follow-up

SECONDARY OUTCOMES:
Improved congruence about end-of-life care between adolescents and family, using the Statement of Treatment Preferences | Measured immediately post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Maureen E. Lyon, PhD, Principal Investigator — Children's Research Institute and Children's National Medical Center
Locations (1):
- Children's Research Institute, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Lyon ME, Garvie PA, Briggs L, He J, McCarter R, D'Angelo LJ. Development, feasibility, and acceptability of the Family/Adolescent-Centered (FACE) Advance Care Planning intervention for adolescents with HIV. J Palliat Med. 2009 Apr;12(4):363-72. doi: 10.1089/jpm.2008.0261. PMID 19327074
- [Background] Lyon ME, Garvie PA, Briggs L, He J, Malow R, D'Angelo LJ, McCarter R. Is it safe? Talking to teens with HIV/AIDS about death and dying: a 3-month evaluation of Family Centered Advance Care (FACE) planning - anxiety, depression, quality of life. HIV AIDS (Auckl). 2010;2:27-37. doi: 10.2147/hiv.s7507. Epub 2010 Feb 18. PMID 22096382
- [Background] Garvie PA, He J, Wang J, D'Angelo LJ, Lyon ME. An exploratory survey of end-of-life attitudes, beliefs, and experiences of adolescents with HIV/AIDS and their families. J Pain Symptom Manage. 2012 Sep;44(3):373-85.e29. doi: 10.1016/j.jpainsymman.2011.09.022. Epub 2012 Jul 7. PMID 22771129
- [Background] Lyon ME, Garvie P, He J, Malow R, McCarter R, D'Angelo LJ. Spiritual well-being among HIV-infected adolescents and their families. J Relig Health. 2014 Jun;53(3):637-53. doi: 10.1007/s10943-012-9657-y. PMID 23104266
- [Result] Lyon ME, Garvie PA, McCarter R, Briggs L, He J, D'Angelo LJ. Who will speak for me? Improving end-of-life decision-making for adolescents with HIV and their families. Pediatrics. 2009 Feb;123(2):e199-206. doi: 10.1542/peds.2008-2379. PMID 19171571